CLINICAL TRIAL: NCT06089837
Title: A Phase 1b Multiple Ascending Dose (MAD) Study of EC5026 in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of Multiple Doses of Oral EC5026 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EicOsis Human Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC5026-1-02
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — EC5026

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EC5026 (Experimental): Multiple Ascending Doses of oral EC5026
  Interventions: Drug: EC5026 oral tablet
- Placebo (Experimental): Single doses of matching oral placebo
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: EC5026 oral tablet — 2 sequential cohorts of 8 subjects randomly assigned to receive multiple ascending oral doses of EC5026 (n=6 per cohort) or matching placebo (n=2 per cohort) for 7 consecutive days.
  Oral doses of EC5026 tested in each cohort:
  4 mg loading dose on Day 1 / 2 mg Maintenance dose on Days 2-7 (Cohort 1) 8 mg loading dose on Day 1 / 4 mg Maintenance dose on Days 2-7 (Cohort 2)
  Arms: EC5026
Drug: Placebo oral tablet — 2 sequential cohorts of 8 subjects randomly assigned to receive multiple ascending oral doses of EC5026 (n=6 per cohort) or matching placebo (n=2 per cohort) for 7 consecutive days. Subject assigned to the Placebo Arm will receive 7 days of matching placebo oral tablets in each Cohort.
  Arms: Placebo

SUMMARY:
EC5026 has been shown to be effective in preclinical pain models of pain, including inflammatory and neuropathic pain subtypes. Two Phase 1a studies - a Phase 1a single ascending dose (SAD) study and a Phase 1a fed-fasted study - have been conducted, evaluating the safety, tolerability, PK, and food effects of single oral doses of EC5026 ranging 0.5 to 24 mg. The present study will evaluate the safety, tolerability, and PK of 2 sequential ascending dose regimens of EC5026, administered once daily for 7 consecutive days, in healthy volunteers.

DETAILED DESCRIPTION:
This is double-blind, randomized, placebo-controlled Phase 1b multiple ascending dose (MAD) study to investigate the safety, tolerability, and pharmacokinetics (PK) of 2 sequential dose regimens of oral EC5026 in healthy male and female subjects.

EC5026 is an inhibitor of the soluble Epoxide Hydrolase (sEH) enzyme developed as a first-in-class analgesic for the treatment of pain. sEH is an enzyme that is downstream in the cytochrome P450 (CYP) pathway of the arachidonic acid (AA) cascade. The sEH enzyme is responsible of metabolizing a class of epoxy-fatty acids known as epoxyeicosatrienoic acids (EETs), which are potent, naturally occurring analgesics. EETs are produced at high concentrations in areas of tissue damage and inflammation, but are rapidly metabolized by the sEH enzyme into inactive compounds. Effective inhibition of sEH activity prolongs the ability of EETs to exert their analgesic activity.

This Phase 1b MAD study will be enrolling 16 healthy male and female subjects 18 years and older. EC5026 and placebo will be administered orally in tablets. Study drug (active or placebo) will be administered as a single oral dose daily, for 7 consecutive days. Subjects assigned to the active drug will receive a single loading dose on Day 1 and a single maintenance dose on Days 2-7. The dose regimens to be assessed in this Phase 1b trial correspond to the following loading dose and maintenance dose pairs: 4 mg/2 mg (Cohort 1, total cumulative 7-day oral dose of 16 mg), and 8 mg/4 mg (Cohort 2, total cumulative 7-day oral dose of 32 mg).

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be enrolled in this study:

1. Male and female subjects must be 18 years or older.
2. Subjects must be willing to provide written informed consent to participate in the study.
3. Subjects must be in generally good health as determined by pre-study medical history, physical examination, clinical laboratory tests, and 12 lead ECG measurements.
4. Subjects must be willing to remain in confinement at the clinical study unit for up to 8.5 consecutive days and to return to the unit as specified for additional blood tests and safety evaluations during the study period.
5. Subjects must have a body mass index (BMI) of 19-32 kg/m2. Participants with a BMI below 19 kg/m2 may be enrolled at the Investigator's discretion.
6. Subjects must have a systolic blood pressure (BP) of 90-160 mmHg, diastolic BP of 50-90 mmHg, and resting HR of 40-100 beats per min without medication at Screening.
7. Subjects must have clinical chemistry values for electrolytes, alkaline phosphatase (ALP), alanine aminotransferase (ALT <1.5x ULN), aspartate aminotransferase (AST, <1.5x ULN), lactate dehydrogenase (LDH), creatine phosphokinase (CPK), creatinine, bilirubin (<2x ULN), and urea that are within the normal range without medication or not clinically significant for a healthy population in the opinion of the Investigator at Screening. Renal clearance measured by eGFR must be normal (≥80 mL/min). Urinalysis values must be within normal limits or not clinically significant for a healthy population in the opinion of the Investigator at Screening. Laboratory analyses and urinalysis may be repeated once at the Investigator's discretion to confirm the accuracy of the results.
8. Subjects must have an early morning (drawn seated between 0600 am and 0800 am) serum cortisol level >5 mcg/dL (>137.9 nmol/L) and early morning adrenocorticotropic hormone (ACTH) and aldosterone levels within the normal range at screening. Randomization will be conditional to a normal cortisol response to ACTH stimulation during screening [serum cortisol level ≥16 mcg/dL (≥440 nmol/L) after IM ACTH injection].
9. Subjects must be non-smokers or previous smokers who have not smoked within the previous 6 months prior to Screening.
10. Male participants must use, from randomization until at least 2 months after the last dose, a highly effective contraception method (less than 1 pregnancy per 100 people using the method for one year), e.g.: sterilisation (e.g., vasectomy), and/or barrier forms of contraception, including condoms (external or internal) and diaphragm ('cap').
11. Male subjects must not donate sperm during the study and for 12 months after receiving the last dose of study drug.
12. Female subjects must be non-pregnant, non-lactating, and either postmenopausal for at least 1 year, or surgically sterile (bilateral tubal ligation ('clipping or tying tubes' or hysterectomy) for at least 3 months, or they must agree to use a highly effective contraception method (less than 1 pregnancy per 100 people using the method for one year), from 28 days and/or their last confirmed menstrual period prior to study enrollment (whichever is longer) until 2 months after clinic discharge. Highly effective contraception methods include: Intra-uterine device (IUD) containing either copper or levonorgestrel (e.g., Mirena®), and/or barrier methods of contraception, including condoms (external or internal) and diaphragm ('cap'). Hormonal methods of contraception (with the exception of hormonal IUD) are not permitted within this study. Female participants will refrain from using hormonal contraceptives for at least 28 days prior to study entry until the end of the study period. Participants/Participant's partner(s) must also use a barrier form of contraception, from the first dose of study drug through until 2 months after the last dose. For all females of childbearing potential, the pregnancy test result must be negative at Screening and Pre-Study Baseline (Day -1).

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Subjects who have used any non-study medication(s), including low-dose aspirin for cardiovascular prophylaxis, within 1 week before administration of study drug.
2. Subjects who have used chemotherapy agents, or who have a personal history of cancer or metastatic cancer in first degree relatives suggestive of elevated cancer risk in the opinion of the investigator, other than nonmetastatic skin cancer that has been completely excised, within 5 years prior to Screening.
3. Subjects with a history of bacterial, fungal, or viral infection requiring treatment with antibiotics, antifungal agents, or antivirals within 1 month prior to randomization.
4. Subjects with a presence or history of peripheral edema within the past 5 years, with the exception of that caused by trauma.
5. Subjects with a history of disorders of the HPA or HPG axis.
6. Subjects with a history of congestive heart failure.
7. Subjects who have used (within 30 days of randomization) or plan on using during the duration of the study any prescription or over-the-counter drugs that are cytochrome P450 (CYP450) inducers or inhibitors (e.g., cimetidine, paroxetine, fluoxetine, haloperidol, ketoconazole, itraconazole, fluconazole, erythromycin, or clarithromycin).
8. Subjects who have used (within 30 days of randomization) or plan on using during the duration of the study any dietary aids, supplements, or foods that are known to modulate drug metabolizing enzymes (e.g., St. John's wort, grapefruit juice).
9. Subjects with difficulty in swallowing oral medications.
10. Subjects with serious psychosocial comorbidities as determined by the Investigator.
11. Subjects with current cognitive or major psychiatric disorders, or any other condition that could interfere with compliance with study procedures and/or confinement in a clinical study unit for up to 8.5 days.
12. Subjects with a positive drug or alcohol test during Screening and/or admission (a positive THC test will be allowed as long as it consists of minimal social use, per discretion of Investigator).
13. Subjects who have used any other investigational drug within 1 month prior to Screening.
14. Subjects who have used any over-the-counter medications within 2 weeks of randomization, or paracetamol or ibuprofen within 7 days of randomization
15. Subjects who have donated and/or received any blood or blood products (more than 450 mL) within 3 months prior to randomization.
16. Subjects with a presence or history of active gastrointestinal disorder, including esophageal or gastroduodenal ulceration, or renal, hepatic, or coagulant disorder within 1 month prior to enrollment.
17. Subjects with a family history of significant cardiac disease (i.e., sudden death in first degree relative; myocardial infarction before the age of 50).
18. Subjects with a cumulative exposure to any oral or inhaled glucocorticoid of more than 1 week duration within 6 months prior to randomization.
19. Subjects with confirmed COVID-19, or suspected COVID-19 (e.g., developed symptoms of a respiratory infection such as cough, sore throat, shortness of breath, or fever, but did not get tested for COVID-19) at the time of Screening.
20. Subjects with confirmed moderate-severe COVID-19 within 2 months of randomization or with confirmed asymptomatic or mild COVID-19 within 4 weeks of randomization.
21. Subjects who have received a COVID-19 vaccine within 4 weeks of randomization or are planning on receiving it during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-05-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAE) [Safety and Tolerability] | 30 days
  All AEs reported or observed during the study will be recorded on the electronic case report forms (eCRF). Information to be collected includes drug treatment, type of event, time of onset, dosage, investigator-specified assessment of severity and relationship to study drug, time of resolution of the event, seriousness, any required treatment or evaluations, and outcome. Any AEs resulting from concurrent illnesses, reactions to concurrent illnesses, reactions to concurrent medications, or progression of disease states must also be reported. All AEs will be followed until they are resolved, stable, or judged by the investigator to be not clinically significant. The Medical Dictionary for Regulatory Activities will be used to code all AEs.
Dose-related effects on electrocardiographic QTc interval (concentration QTc analysis) | 7 days
  Study participants will be wearing a ECG-Holter monitoring during the 7 days of dosing with study drug (EC5026 or placebo). ECG extractions will be performed concurrently with PK timepoints for concentration QTc analysis.
Changes-from-baseline in electrocardiographic time intervals | 7 days
  Study participants will be wearing a ECG-Holter monitoring during the 7 days of dosing with study drug (EC5026 or placebo). ECG extractions will be performed concurrently with PK timepoints. Assessments will include evaluating changes-from-baseline heart rate (HR), PR interval, QRS interval, and QTc interval within the Holter ECG recording. All intervals are measured in time (msec).
Area under the plasma concentration versus time curve (AUC) in response to 2 multiple ascending dose regimens of EC5026 oral tablets [Plasma Pharmacokinetics]. | 30 days
  Standard noncompartmental methods will be used.
Maximum observed plasma concentration (Cmax) in response to 2 multiple ascending dose regimens of EC5026 oral tablets [Plasma Pharmacokinetics]. | 30 days
  Standard noncompartmental methods will be used.
Time to maximum observed plasma concentration (Tmax) in response to 2 multiple ascending dose regimens of EC5026 oral tablets [Plasma Pharmacokinetics]. | 30 days
  Standard noncompartmental methods will be used.
Terminal elimination rate constant in plasma (Kel) in response to 2 multiple ascending dose regimens of EC5026 oral tablets [Plasma Pharmacokinetics]. | 30 days
  Standard noncompartmental methods will be used.
Terminal phase half-life in plasma (t1/2) in response to 2 multiple ascending dose regimens of EC5026 oral tablets [Plasma Pharmacokinetics]. | 30 days
  Standard noncompartmental methods will be used.
Apparent total body clearance (CL/F) in response to 2 multiple ascending dose regimens of EC5026 oral tablets [Plasma Pharmacokinetics]. | 30 days
  Standard noncompartmental methods will be used.
Apparent volume of distribution based on the terminal elimination rate constant in plasma (Vz/F) in response to 2 multiple ascending dose regimens of EC5026 oral tablets [Plasma Pharmacokinetics]. | 30 days
  Standard noncompartmental methods will be used.
Renal clearance (CLR) in response to 2 multiple ascending dose regimens of EC5026 oral tablets [Plasma Pharmacokinetics]. | 7 days
  Standard noncompartmental methods will be used.
Amount of drug excreted unchanged in urine (Ae) in response to 2 multiple ascending dose regimens of EC5026 oral tablets [Plasma Pharmacokinetics]. | 7 days
  Standard noncompartmental methods will be used.
Fraction of eliminated dose in urine (Fe%) in response to 2 multiple ascending dose regimens of EC5026 oral tablets [Plasma Pharmacokinetics]. | 7 days
  Standard noncompartmental methods will be used.

OTHER OUTCOMES:
Effects of 2 ascending multiple dose regimens of EC5026 versus placebo on oxylipin biomarkers. | 30 days
  Standard validated oxylipin measurement platform will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Cory D Sellwood, MBChB, Principal Investigator — New Zealand Clinical Research; William K Schmidt, PhD, Study Director — EicOsis Human Health Inc.
Locations (1):
- New Zealand Clinical Research, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No